CLINICAL TRIAL: NCT04082962
Title: Dexamethasone Intravitreal Implant for the Management of Exudative Retinal Detachment in Patients With Uveal Melanoma
Brief Title: Dexamethasone Implant for Retinal Detachment in Uveal Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ivana K. Kim (Other)
Responsible Party: Sponsor-Investigator, Ivana K. Kim, Associate Professor of Ophthalmology, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019P000127
Record Dates: First submitted 2019-08-27; First posted 2019-09-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Exudative Retinal Detachment and Uveal Melanoma
Keywords: Dexamethasone; Uveal Melanoma; Steroid-Implant; Exudative Retinal Detachment
MeSH Terms: conditions — Uveal Melanoma | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Twenty patients will be enrolled in this randomized pilot study. Patients will be randomized (1:1) to receive the dexamethasone implant or no treatment. A stratified randomization scheme will be performed, with strata defined by tumor height (< 5mm and 5mm - < 10 mm). Patients with newly diagnosed choroidal melanoma meeting specified eligibility criteria will be randomly assigned to receive Ozurdex™ (0.7 mg dexamethasone) or no treatment at the time of their tumor localization (tantalum ring placement) surgery for patients receiving PBI or at the time of plaque removal for those patients receiving plaque radiotherapy.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Participants receiving dexamethasone implant.
  Interventions: Drug: Dexamethasone intravitreal implant
- Non-treatment group (control) (No Intervention): Participants not receiving dexamethasone implant.

INTERVENTIONS:
Drug: Dexamethasone intravitreal implant — Ozurdex™ is an intravitreal implant containing dexamethasone 0.7 mg in the NOVADUR® solid polymer drug delivery system (NOVADUR™ system contains poly (D,L-lactide-co-glycolide) PLGA intravitreal polymer matrix, which slowly degrades to lactic acid and glycolic acid.). Ozurdex™ is preservative-free. It is supplied in a foil pouch with a single-use plastic applicator.
  Other Names: Ozurdex™
  Arms: Treatment Group

SUMMARY:
This is an investigator-initiated Phase I study of a single dose of an intravitreally-administered dexamethasone implant (Ozurdex™) in subjects with uveal melanomas (UM) and exudative retinal detachments (ERD: build-up of fluid under the retina that causes it to detach) being treated with proton beam radiation (PBI) or plaque radiotherapy. Although PBI is an effective treatment for UM, ERDs may persist after radiation, leading to vision loss. Effective treatments for ERD are currently lacking. We are conducting this study to evaluate whether Ozurdex™ can help resolve ERDs that occur in patients with UM. Ozurdex™ has been approved by the Food and Drug Administration (FDA) to treat certain ocular conditions such as macular edema, non-infectious uveitis, and diabetic macular edema but it is not approved for use in patients with UM and ERD. This study will determine the safety of the dexamethasone implant and provide preliminary evidence of efficacy in this population.

DETAILED DESCRIPTION:
Study Objective: The primary objective of the study will be to determine the safety of the Ozurdex (dexamethasone) intravitreal implant. The secondary objective is to determine if the implant helps to resolve exudative retinal detachment, a secondary complication associated with uveal melanoma.

Background: This is a single site investigator-initiated Phase I study of a single dose of intravitreally administered dexamethasone implant (Ozurdex™) in subjects with choroidal melanomas and exudative retinal detachments being treated with proton beam irradiation or plaque radiation therapy. This is one of the first studies to evaluate the Ozurdex™ implant in this setting. Therefore the primary goal is to evaluate safety.

Patient Population: Twenty patients will be enrolled in this randomized pilot study. Patients must meet the following eligibility criteria to enroll: Tumor thickness ≤ 10 mm, associated serous retinal detachment > two clock hours in extent, primary treatment of ocular melanoma with proton irradiation or plaque radiotherapy. Males and females >18 years of age are eligible.

Methods: Patients will be randomized (1:1) to receive the dexamethasone implant or no treatment. A stratified randomization scheme will be performed, with strata defined by tumor height (< 5mm and 5mm - ≤ 10 mm). Patients will be masked to their treatment assignment.

Patients will be randomly assigned to receive Ozurdex™ (0.7 mg dexamethasone) or no treatment at either (1) the time of their tumor localization (tantalum ring placement) surgery before proton therapy or (2) their surgery removing the plaque following plaque radiotherapy. A sham treatment procedure to maintain the mask will be unnecessary.

Patients will be followed at 6 weeks, 14 weeks, 28 weeks and 54 weeks after administration of the dexamethasone implant. Visual acuity, intraocular pressure, optical coherence tomography, B-scan ultrasonography, wide-angle color photography and full ophthalmological examination will be performed pre-op and on every follow-up visit. Evaluation of adverse events and review of medical history and medication use will be completed at all follow-up visits.

The primary outcome of the study will be to evaluate the safety of the implant. This will be done by monitoring for all adverse effects not related to the melanoma or radiation treatment including significant vision loss, other sight-threatening events, and unforeseen systemic events.

Secondary endpoints include resolution of retinal detachment at 6 and 12 months after implant insertion, visual acuity at 6 and 12 months after implant insertion, and development of iris neovascularization and neovascular glaucoma during the 12 month study period.

Statistical Analysis Plan: There is no formal sample size calculation in a pilot/phase I study. As this is a phase I study, a sample size of 20 patients is chosen, making sure that it is feasible financially and logistically to conduct the study.

Safety Endpoints: Incidence and severity of ocular and systemic adverse events identified by ocular examination, diagnostic tests, and subject reporting will be summarized. Comparisons of these endpoints of study subjects who received treatment may be made with those of control subjects, matched on prognostic factors including tumor size and tumor location. The proportion of treated patients with adverse events will be tabulated by body system, stratified by tumor size and location, and compared to patients in the control arm using Fisher's exact test and other appropriate tests of association.

Efficacy Endpoints: Descriptive statistics will be generated to assess resolution of exudative retinal detachment at 6 months after placement of the Ozurdex implant or no treatment. This is the most important efficacy endpoint. Descriptive statistics will be generated for the following secondary efficacy endpoints: incidence of neovascular glaucoma, incidence of rubeosis, percent of patients with exudative retinal detachment at 12 months, and distribution of visual acuity measures at 6 months and 12 months. All measures will be compared between patients in the treatment arm and those in the control arm of the study.

ELIGIBILITY:
Inclusion Criteria:

* Tumor thickness <= 10 mm.
* Associated serous retinal detachment extending beyond tumor, > two clockhours in extent.
* Primary treatment of ocular melanoma with proton irradiation or plaque radiotherapy.

Exclusion Criteria:

* Any pre-existing glaucoma.
* History of elevated IOP (> 25 mm Hg).
* History of steroid response glaucoma.
* Active or suspected ocular or periocular infections including most viral diseases of the cornea and conjunctiva: active ocular herpes simplex, active epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, varicella, mycobacterial infections, and fungal diseases.
* Any history of ocular herpes simplex.
* Torn or ruptured posterior lens capsule.
* Known hypersensitivity to any components of the dexamethasone intravitreal implant.
* Women of child-bearing potential: pregnant or planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events Related to the Implant | Throughout 12 month study period
  The primary outcome of the study will be to evaluate the safety of the implant. All adverse effects not related to the melanoma or radiation treatment identified by ocular examination, diagnostic tests, and subject reporting will be tabulated. This includes significant vision loss, other sight-threatening events, and unforeseen systemic events.

SECONDARY OUTCOMES:
Exudative retinal detachment resolution | 6 and 12 months after implant insertion
  Will be assessed using spectral domain optical coherence tomography, B-scan ultrasonography, and Optos wide-angle color photography.
Visual Acuity | 6 and 12 months after implant insertion
  Measured with ETDRS chart.
Complications | Throughout 12 month study period.
  The development of iris neovascularization and neovascular glaucoma.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana K Kim, MD, Principal Investigator — Harvard Medical School, Massachusetts Eye and Ear
Locations (1):
- Anne Marie Lane, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scotto J, Fraumeni JF Jr, Lee JA. Melanomas of the eye and other noncutaneous sites: epidemiologic aspects. J Natl Cancer Inst. 1976 Mar;56(3):489-91. doi: 10.1093/jnci/56.3.489. PMID 1255781
- [Background] Collaborative Ocular Melanoma Study Group. The COMS randomized trial of iodine 125 brachytherapy for choroidal melanoma: V. Twelve-year mortality rates and prognostic factors: COMS report No. 28. Arch Ophthalmol. 2006 Dec;124(12):1684-93. doi: 10.1001/archopht.124.12.1684. PMID 17159027
- [Background] Gragoudas ES. Proton beam irradiation of uveal melanomas: the first 30 years. The Weisenfeld Lecture. Invest Ophthalmol Vis Sci. 2006 Nov;47(11):4666-73. doi: 10.1167/iovs.06-0659. No abstract available. PMID 17065472
- [Background] Kivela T, Eskelin S, Makitie T, Summanen P. Exudative retinal detachment from malignant uveal melanoma: predictors and prognostic significance. Invest Ophthalmol Vis Sci. 2001 Aug;42(9):2085-93. PMID 11481276
- [Background] Gibran SK, Kapoor KG. Management of exudative retinal detachment in choroidal melanoma. Clin Exp Ophthalmol. 2009 Sep;37(7):654-9. doi: 10.1111/j.1442-9071.2009.02127.x. PMID 19788660
- [Background] Char DH, Bove R, Phillips TL. Laser and proton radiation to reduce uveal melanoma-associated exudative retinal detachments. Am J Ophthalmol. 2003 Jul;136(1):180-2. PMID 12834689
- [Background] Parrozzani R, Pilotto E, Dario A, Miglionico G, Midena E. Intravitreal triamcinolone versus intravitreal bevacizumab in the treatment of exudative retinal detachment secondary to posterior uveal melanoma. Am J Ophthalmol. 2013 Jan;155(1):127-133.e2. doi: 10.1016/j.ajo.2012.06.026. Epub 2012 Sep 18. PMID 22995029
- [Background] Kim IK, Lane AM, Jain P, Awh C, Gragoudas ES. Ranibizumab for the Prevention of Radiation Complications in Patients Treated With Proton Beam Irradiation for Choroidal Melanoma. Trans Am Ophthalmol Soc. 2016 Aug;114:T2. PMID 27630373
- [Background] Malcles A, Nguyen AM, Mathis T, Grange JD, Kodjikian L. Intravitreal dexamethasone implant (Ozurdex(R)) for exudative retinal detachment after proton beam therapy for choroidal melanoma. Eur J Ophthalmol. 2017 Aug 30;27(5):596-600. doi: 10.5301/ejo.5000940. Epub 2017 Feb 8. PMID 28218368
- [Background] Koehler PJ. Use of corticosteroids in neuro-oncology. Anticancer Drugs. 1995 Feb;6(1):19-33. doi: 10.1097/00001813-199502000-00002. PMID 7756680
- [Background] Sturdza A, Millar BA, Bana N, Laperriere N, Pond G, Wong RK, Bezjak A. The use and toxicity of steroids in the management of patients with brain metastases. Support Care Cancer. 2008 Sep;16(9):1041-8. doi: 10.1007/s00520-007-0395-8. Epub 2008 Feb 7. PMID 18256860